CLINICAL TRIAL: NCT00678236
Title: A Migration and Bone Density Study Comparing Refobacin Bone Cement R vs. Refobacin Plus Bone Cement in the OptiPac Bone Cement Mixing System. A Prospective Randomized Study on Primary Total Knee Arthroplasty
Brief Title: A Migration and Bone Density Study Comparing 2 Types of Bone Cement in the OptiPac Bone Cement Mixing System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 20070237
Record Dates: First submitted 2008-05-08; First posted 2008-05-15 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Osteoarthritis
Keywords: RSA; Gonarthritis; Bone Cement
MeSH Terms: conditions — Osteoarthritis | interventions — gentamicin-polymethylmethacrylate bead; Bone Cements

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Refobacin Bone Cement R
  Interventions: Other: Refobacin Bone Cement R
- 2 (Active Comparator): Refobacin Plus Bone Cement
  Interventions: Other: Refobacin Plus Bone Cement

INTERVENTIONS:
Other: Refobacin Bone Cement R — Insertion of a knee prosthesis fixed by Refobacin Bone Cement R
  Other Names: Biomet Europe: Refobacin Bone Cement R
  Arms: 1
Other: Refobacin Plus Bone Cement — Insertion of a knee prosthesis fixed by Refobacin Plus Bone Cement
  Other Names: Biomet Europe: Refobacin Plus Bone Cement
  Arms: 2

SUMMARY:
The goal of this scientific study is to determine whether there are differences in early migration and prosthesis-near bone density when a standard knee prosthesis is fixed with Refobacin Bone Cement R or with Refobacin Plus Bone Cement. Migration will be evaluated with RSA and bone density around the prosthesis with DEXA. The study will be successful if the prosthesis is fixed and remains in place throughout the entire period of the study, that is, that there is no increasing migration as measured by RSA. The cement type that ensures the largest number of solidly fixed prostheses during the two-year evaluation period will be "the best".

DETAILED DESCRIPTION:
Loosening of prosthetic components continues to play a large role in total knee alloplasty (TKA) and need for revision. Osteolysis is an important part of prosthesis loosening, but we still do not completely understand the mechanism. Research has shown that mechanical factors such as weak bone cement and poor contact between cement/bone or cement/implant interphase contribute to loosening of implants. Survival of cemented TKA components also depend on a careful balancing of soft tissues around the knee, repair of lower extremity dislocations, design of the prosthesis and the level of patients' activities. Sclerosis of the proximal tibia can present a problem with regard to getting the cement to penetrate into the bone. Poor operative technique, such as high volume or high pressure lavage of the prepared bone surface, can result in reduced penetration of cement into the spongiosa and early failure of the prosthesis, measured as progressive radiolucent lines (RLLs). En tourniquet counter acts bleeding at the implant site and provides for better penetration of cement into the trabeculae of the bone. If the bone surface at the implantation site is contaminated with blood before the cement is applied, the shear strength in the bone/cement interphase can be reduced by up to 50%.

In prosthesis used in this study includes a tibial plateau with a central stem with stabilizing wings, the bottom surface of which is recessed by about 1 mm, so that a pocket is formed surrounded by a lip that provides for an even thickness of the cement layer beneath the tibial plateau. This assures that the cement is pressed down into the spongiosa during fixation of the implant. This design doubles the penetration of the cement compared with prostheses without a depressed baseplate. The company behind this design has had a successful follow-up of this system for more than 15 years. A good cement/implant interphase lessens the risk of penetration of debris into the interphase and thus reduces the risk for the development of osteolysis and aseptic loosening of the implant.

Fixation of knee alloplasties is done in 70% of cases with use of cement. It is uncertain whether there is a difference in the long-term survival of knee prostheses with the two types of cement used in this project. Both types of cement in this study are used today in knee surgery with good, short-term clinical results. It is important to investigate new types of cement in order to assure future patients the best possible results after knee alloplasty and fewer re-operations.

The goal of this scientific study is to determine whether there are differences in early migration and prosthesis-near bone density when a standard knee prosthesis is fixed with Refobacin Bone Cement R or with Refobacin Plus Bone Cement. Migration will be evaluated with RSA and bone density around the prosthesis with DEXA. The study will be successful if the prosthesis is fixed and remains in place throughout the entire period of the study, that is, that there is no increasing migration as measured by RSA. The cement type that ensures the largest number of solidly fixed prostheses during the two-year evaluation period will be "the best".

ELIGIBILITY:
Inclusion Criteria:

* primary or secondary knee osteoarthritis
* sufficient bone quality for total knee arthroplasty
* age above 70 years
* no upper age limit if the patient is capable
* informed and written consent
* patient can only enter the project with one knee

Exclusion Criteria:

* neuromuscular or vascular disease in the affected leg
* preoperatively not found suitable for a knee arthroplasty
* patients with osteoporosis based on former diagnosis or preoperative DEXA-scan
* fracture sequelae or previous PTO or previous extensive knee surgery
* patients with need of a stem-elongation
* patients who cannot refrain from taking NSAID post-operatively
* continuous medical treatment with vitamin K antagonists (Warfarin) which is known to reduce the bon emineral density by a factor of 5
* patients with metabolic bone disease
* patients with rheumatoid arthritis
* postmenopausal women in estrogenic hormone substitution
* patients with a continuous need of systemic cortisone treatment
* non-Danish citizenship
* patients who do not comprehend the Danish language (read and speak)
* senile dementia
* alcoholism - defined as men drinking more than 21 units a week and women drinking more than 14 units a week
* drug abuse
* major psychiatric disease
* metastatic cancer disease and treatment with radiation therapy or chemotherapy
* severe systemic disease (e.g. hemi paresis and Parkinson disease)
* systemic hip and spine disease
* employee at the orthopaedic department, Aarhus University Hospital
* ongoing case regarding industrial injury insurance of the knee
* patients with poor dental status (risk of infection)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Tibial implant migration evaluated by RSA | 2013

SECONDARY OUTCOMES:
Comparison of Refobacin Bone Cement R vs. Refobacin Plus Bone Cement | 2013

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Soballe, MD, Prof., Principal Investigator — Orthopaedic Center, Aarhus University Hospital, Tage-Hansens Gade 2, 8000 Århus C, Denmark
Locations (1):
- Orthopaedic Center, Aarhus University Hospital, Aarhus, Denmark